CLINICAL TRIAL: NCT03362086
Title: Establishment of Osteosarcoma Biobank
Brief Title: The Osteosarcoma Biobank in Peking University People's Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ren tingting, Lab manager of Musculoskeletal Tumor Center, Peking University People's Hospital
Other Study IDs: PKU-osteosarcoma
Record Dates: First submitted 2017-11-26; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Osteosarcoma
Keywords: bone tumor osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigator will collect pecimen and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteosarcoma is very rare bone tumor. The investigator set up the biobank to ensure the patients has the chance to participate in future research

DETAILED DESCRIPTION:
Samples of blood and other stored material such as slides,frozen tissues and so on .

Questionnaire information, including health history, growth and development, physical activity and family medical history information.

ELIGIBILITY:
Inclusion Criteria:

Proband Inclusion criteria: A diagnosis or suspected diagnosis of osteosarcoma

Exclusion Criteria:

non-asian pulmonary metastasis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the patients diagnosed with osteosarcoma without pulmonary metastasis
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Examine VEGFR-2 and PD-L1 gene expression osteosarcoma | 3 years
  To examine the VEGFR2 and programmed cell death ligand 1 (PD-L1) genes expression of the patients with osteosarcoma.And Analyze their differences.

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Ren, phD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided